CLINICAL TRIAL: NCT04399863
Title: Feasibility Study of the ETOILE Program, a Therapeutic Education Program in Pediatric Hematology About Acute Lymphoblastic Leukemia and Allogenic Hematopoietic Steam Cells Transplantation, for Patient and Caregivers
Brief Title: ETOILE : A Feasibility Study in Pediatric Patient Education
Acronym: ETOILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP200113; IDRCB: 2019-A03127-50 (Other: French Health Autority)
Record Dates: First submitted 2020-05-11; First posted 2020-05-22 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2020-05

CONDITIONS: Leukemia, Lymphoblastic
Keywords: therapeutic education
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETOILE therapeutic education (Experimental): ETOILE is a patient education program, in accordance with French recommendations, which offers to patients and caregivers the opportunity to follow a customized educational training on their disease. Better quality of life and enhanced autonomy are the aim of this program.
  Interventions: Behavioral: ETOILE therapeutic education

INTERVENTIONS:
Behavioral: ETOILE therapeutic education — ETOILE is a patient education program, in accordance with French recommendations, which offers to patients and caregivers the opportunity to follow a customized educational training on their disease. Better quality of life and enhanced autonomy are the aim of this program.

SUMMARY:
Feasibility study of a therapeutic education program for the patient and his carers, intended for children suffering from acute lymphoblastic leukemia or having received an allograft of hematopoietic stem cells in the pediatric hematology department of Robert Debré hospital ( Paris, APHP). In addition to feasibility, the intermediate effectiveness of the program will be assessed.

DETAILED DESCRIPTION:
This is a pilot feasibility study, of the quasi-experimental before-after, non-randomized, mono-centric type. Feasibility is assessed on process criteria (adoption, reach implementation, satisfaction). Intermediate effectiveness is assessed on the skill level of patients and their caregivers, before, after and at a distance from education. Patients' anxiety levels will also be assessed before, after and at a distance from the program. The level of health literacy will be assessed at the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Criteria relating to the population studied: child between 0 and 18 years old, followed at Robert Debré hospital (Paris), by a doctor from the hematology and immunology department

  * Of which the 2 holders of parental authority have been informed and have signed the consent
  * Having 1 or 2 caregivers available to accompany him during FTE sessions
  * 1 to 2 of their adult caregivers will be eligible for the ETOILE program and will be included in the study after their consent.
  * Child with acute lymphoblastic leukemia, treated at Robert Debré Hospital (Paris), in the induction or consolidation phase
  * Child going to receive or having received an allograft of hematopoietic stem cells at the Robert Debré hospital (Paris)
  * Beneficiaries of a social security scheme or entitled to it,

Exclusion Criteria:

* Child not mastering the French language,
* Child with physical or cognitive disability to participate in the program,

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the ETOILE program | 6 months
  number of patients which joined the programme compared to number of patients referred

CONTACTS AND LOCATIONS:
Overall Officials: Julie ROUPRET-SERZEC, PharmD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No